CLINICAL TRIAL: NCT06032962
Title: Opportunistic Salpingectomy in Non-gynecological Surgeries - a Pilot Study
Brief Title: Opportunistic Salpingectomy in Non-gynecological Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana Josephy (Other)
Responsible Party: Sponsor-Investigator, Dana Josephy, Dana Josephy, Meir Medical Center
Organization: Meir Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MeirMedicalCenter
Record Dates: First submitted 2023-07-19; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer Prevention
MeSH Terms: interventions — Salpingectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-gynecologic surgery (Experimental): Female candidates for non-gynecologic abdominal surgery
  Interventions: Procedure: salpingectomy

INTERVENTIONS:
Procedure: salpingectomy — surgical removal of the fallopian tubes

SUMMARY:
The goal of this study is to evaluate patient's compliance for opportunistic salpingectomy (OS) and procedure feasibility in non gynecological abdominal surgeries

DETAILED DESCRIPTION:
Patients who are candidate for non-gynecological abdominal surgery, are offered OS. If agree, a general surgeon perform the procedure during the planned abdominal surgery

ELIGIBILITY:
Inclusion Criteria:

* Women who were candidates for non-gynecological abdominal surgery
* Aged 45 or older, or aged 40 or older with a desire for bilateral salpingectomy

Exclusion Criteria:

* Pregnant women
* Candidates for urgent surgery

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
patients willing for salpingectomy | day of enrollment
  The number of patients that will agree for salpingectomy
patients undergoing salpingectomy | from enrollment and up to 6 weeks
  The number of patients that will undergo salpingectomy
length of salpingectomy | within surgery
  the length (in minutes) of salpingectomy
surgical complications | up to 30 days from surgery
  complications during or after salpingectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel